CLINICAL TRIAL: NCT05825066
Title: Sequential Neoadjuvant Chemotherapy for Borderline Resectable and Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Neoadjuvant Chemotherapy for Borderline Resectable and Locally Advanced Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00095699; WFBCCC 57222 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pancreas Adenocarcinoma; Borderline Resectable Pancreatic Adenocarcinoma; Locally Advanced Pancreatic Adenocarcinoma
MeSH Terms: interventions — Taxes; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Chemotherapy (Gemcitabine and nab-Paclitaxel and mFOLFIRNIOX) (Experimental): * Gemcitabine (1000 mg/m2 weekly, on day 1,8 and 15 OR 1000 mg/m2 weekly, on day 1 and 15 over 30 minutes after nab-paclitaxel infusion.
  * nab-Paclitaxel (125 mg/m2 weekly, on days 1,8, and 15 OR on days 1 and 15 as a 30-40 minute infusion administered first) for one month and then transition to mFOLFIRNIOX for one month
    1 Cycle = 4 weeks: Day 1,8,15 in a 28 day cycle; 3 consecutive weeks (weeks 1, 2, and 3) of chemotherapy with 1 week off, OR
    1 Cycle = 4 weeks: Day 1, 15 in a 28 day cycle; Every other week (weeks 1 and 3) of chemotherapy with 2nd and 4th week off
  * mFOLFIRINOX: Oxaliplatin, 85 mg/m² IV once every two weeks over 2 hours on Day 1 Irinotecan, 150 mg/m² IV once every two weeks over 90 minutes on Day 1 5-FU, 2,400 mg/m² IV once every two weeks over 46-48 hours administered via infusion Leucovorin, 400 mg/m2 IV every two weeks over 90 minutes on Day 1
    1. Cycle = 4 weeks, administration on Day 1 and Day 15 of each mFOLIRINOX cycle
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Other: Radiological Assessments; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Nab paclitaxel — The intervention will be administered on an outpatient basis. The patients on this study will begin treatment with GA for one month and then transition to mFFX for one month.
  The patient will come off of the sequence study intervention if the imaging after the 2nd month shows unequivocal progression. After four months of sequential neoadjuvant therapy the patient will come off study and can proceed to surgery, radiation, or extended course of chemotherapy as determined by the multidisciplinary tumor board consensus or the treating physician.
Drug: Gemcitabine — The intervention will be administered on an outpatient basis. The patients on this study will begin treatment with GA for one month and then transition to mFFX for one month.
  The patient will come off of the sequence study intervention if the imaging after the 2nd month shows unequivocal progression. After four months of sequential neoadjuvant therapy the patient will come off study and can proceed to surgery, radiation, or extended course of chemotherapy as determined by the multidisciplinary tumor board consensus or the treating physician.
Other: Radiological Assessments — CT imaging of chest abdomen and pelvis will be performed every 8 weeks. MRI may be used.
Drug: mFOLFIRINOX — The intervention will be administered on an outpatient basis. The patients on this study will begin treatment with GA for one month and then transition to mFFX for one month.
  The patient will come off of the sequence study intervention if the imaging after the 2nd month shows unequivocal progression. After four months of sequential neoadjuvant therapy the patient will come off study and can proceed to surgery, radiation, or extended course of chemotherapy as determined by the multidisciplinary tumor board consensus or the treating physician.

SUMMARY:
The objective of this research is to find out what effects (good and bad), the sequence of Gemcitabine - Abraxane (nab-Paclitaxel) followed by mFOLFIRINOX, the standard chemotherapy for pancreatic cancer, has on participants and their condition. Gemcitabine - Abraxane (nab-Paclitaxel) and mFOLFIRINOX has been approved by the US Food and Drug Administration (FDA) as first line treatment for advanced pancreatic cancer. The sequence of Gemcitabine - Abraxane (nab-Paclitaxel) followed by mFOLFIRINOX has not been approved by the FDA for treatment of pancreatic cancer.

DETAILED DESCRIPTION:
Primary Objective:

- The primary objective of this study is to evaluate the efficacy of sequential Gemcitabine - Abraxane (nab-Paclitaxel) followed by mFOLFIRINOX in improving R0 resection rate in patients with borderline resectable pancreatic cancer and locally advanced unresectable pancreatic cancer.

Secondary Objectives:

* Evaluate the safety and tolerability of sequential Gemcitabine - Abraxane (nab-Paclitaxel) followed by mFOLFIRINOX in patients with borderline resectable pancreatic cancer and locally advanced unresectable pancreatic cancer
* Evaluate progression-free survival (PFS) in patients treated with sequential Gemcitabine - Abraxane (nab-Paclitaxel) followed by mFOLFIRINOX in patients with borderline resectable pancreatic cancer and locally advanced unresectable pancreatic cancer according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) guidelines
* Evaluate overall survival (OS) in patients treated with sequential Gemcitabine - Abraxane (nab-Paclitaxel) followed by mFOLFIRINOX in patients with borderline resectable pancreatic cancer and locally advanced unresectable pancreatic cancer
* Evaluate the objective response rate (ORR) in patients treated with sequential Gemcitabine - Abraxane (nab-Paclitaxel) followed by mFOLFIRINOX in patients with borderline resectable pancreatic cancer and locally advanced unresectable pancreatic cancer.
* Evaluate the disease control rate (DCR) in patients treated with Gemcitabine - Abraxane (nab-Paclitaxel) followed by mFOLFIRINOX in patients with borderline resectable pancreatic cancer and locally advanced unresectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven adenocarcinoma of the pancreas. Patients with mixed tumor with predominant adenocarcinoma pathology can be enrolled
* Patients with borderline resectable or locally advanced pancreatic adenocarcinoma as assessed per NCCN guidelines (either pancreatic head, neck, uncinate process, or body/tail) or institutional multidisciplinary consensus
* Age 18 or above
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Patients must have organ and marrow function as defined below:

Hemoglobin* ≥8 g/dL Absolute neutrophil count ≥1,500/mcL Platelets* ≥100,000/mcL Total bilirubin* ≤1.5 X institutional upper limit of normal AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal Creatinine ≤1.5 X institutional upper limit of normal or CrCL>50

* It is acceptable to transfuse packed red blood cells (PRBC) and platelets at the time of enrollment to meet the eligibility criteria.
* If obstructive jaundice is present, consider ursodiol or a biliary drainage procedure. If the total bilirubin can be reduced or kept to less than or equal to 3 mg/dL, then this inclusion criteria is met.

  * Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
  * Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative)

Exclusion Criteria:

* Patients who have had prior chemotherapy with gemcitabine and/or nab-paclitaxel or FOLFIRINOX for pancreatic cancer
* Patients receiving any other investigational anti-neoplastic agents
* History of malignancy in last 3 years except cervical cancer in situ, adequately treated basal cell or squamous cell carcinoma of skin or treated low risk prostate cancer, who are considered to be eligible
* Patients with active and uncontrolled bacterial, viral or fungal infection requiring systemic therapy. Patients can be reevaluated for the study if the infection is deemed to be under control and the systemic therapy for the infection is completed
* Uncontrolled intercurrent illness including, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the patient's safety
* Patients with known diagnosis of interstitial lung disease, sarcoidosis, pulmonary fibrosis, or pneumonitis requiring oxygen supplementation. Those that do not require oxygen supplementation are eligible.
* Patients who have undergone surgery, other than diagnostic or minor procedures, within 4 weeks prior to the initiation of study treatment
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate - Borderline Resectable Prostate Cancer Participants | 9 months
  The R0 resection is assessed only in patients who undergo surgery. R0 resection is a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed. Participants are considered to be evaluable if they receive at least one sequence of treatments with GA and mFFX (1 cycle GA followed by 1 cycle of m FFX). Primary analysis for each cohort will calculate the R0 resection rate with one-sided 95% confidence interval.
R0 Resection Rate - Locally Advanced Prostate Cancer Participants | 9 months
  The R0 resection is assessed only in patients who undergo surgery. R0 resection is a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed. Participants are considered to be evaluable if they receive at least one sequence of treatments with GA and mFFX (1 cycle GA followed by 1 cycle of m FFX). Primary analysis for each cohort will calculate the R0 resection rate with one-sided 95% confidence interval.

SECONDARY OUTCOMES:
Incidences of Adverse Events | Up to 1 year after completion of study intervention
  The incidence of treatment-emergent toxicities/adverse events (AEs) and Serious Adverse Events (SAEs) in terms categorized and graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5). Incidence tables will be generated to summarize incidence of patients reporting at least one episode of each specific adverse event, incidence of adverse events causing withdrawals and incidence of serious adverse events, separated by cohort.
Number of Participants to Complete Study Intervention | 9 months
  The number of participants to complete 4 cycles of sequential chemotherapy.
Progression-Free Survival (PFS) | Up to 1 year after completion of study intervention
  Progression free survival (PFS) is defined from the day of study treatment initiation until progression according to RECIST v 1.1 guidelines (d. Progression: One or more of the following must occur: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, as well as an absolute increase of at least 0.5 cm. Unequivocal progression of non-measurable disease in the opinion of the treating physician) or death of any cause, whichever occurs first, as measured throughout the study. Stratified Kaplan-Meier curves will be constructed to assess PFS with estimated 6-month and median times with 95% confidence intervals
Overall Survival (OS) | Up to 1 year after completion of study intervention
  Overall survival (OS) is defined from the time of study treatment initiation until death of any cause. Stratified Kaplan-Meier curves will be constructed to assess OS with estimated 6-month and median times with 95% confidence intervals
Tumor Response | Up to 1 year after completion of study intervention
  Tumor response based defined as the proportion of patients who achieve complete response or partial response based on RECISTv1.1 criteria. These will be evaluated according to the RECISTv1.1 criteria using a summarized count/percent with one-sided 95% confidence interval for each cohort:
  The RECIST v1.1 definitions include:
  Complete Response (CR): The disappearance of all target lesions.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
Treatment Response | Up to 1 year after completion of study intervention
  Treatment response is defined as the proportion of patients with a disease control rate (complete + partial response + stable disease) based on RECISTv1.1 criteria using a summarized count/percent with one-sided 95% confidence interval for each cohort.
  Complete Response (CR): Complete disappearance of all target and non-target lesions (with the exception of lymph nodes mentioned below). No new lesions. No disease related symptoms.
  Partial Response (PR): Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions.
  Stable: Does not qualify for CR, PR, Progression or Symptomatic Deterioration. All target measurable lesions must be assessed using the same techniques as baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi K Paluri, MD, MPH, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No